CLINICAL TRIAL: NCT01146210
Title: Identification of de Novo Fanconi Anemia Patients Using FANCD2 Western Blots
Brief Title: Identification of de Novo Fanconi Anemia in Younger Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B2; NCI-2011-02219 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AAML10B2 (Other: Childrens Oncology Group); CDR0000671437 (Other: Clinical Trials.gov); AAML10B2 (Other: Children's Oncology Group); AAML10B2 (Other: CTEP)
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Acute Erythroleukemia (M6); Childhood Acute Megakaryocytic Leukemia (M7); Childhood Acute Minimally Differentiated Myeloid Leukemia (M0); Childhood Acute Monoblastic Leukemia (M5a); Childhood Acute Monocytic Leukemia (M5b); Childhood Acute Myeloblastic Leukemia With Maturation (M2); Childhood Acute Myeloblastic Leukemia Without Maturation (M1); Childhood Acute Myelomonocytic Leukemia (M4); Childhood Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Fanconi Anemia; Refractory Anemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Refractory Anemia With Ringed Sideroblasts; Secondary Myelodysplastic Syndromes; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Fanconi Anemia; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-correlative: Previously collected cryopreserved cells are analyzed via western blot to identify patients with Fanconi anemia.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research study is studying identification of de novo Fanconi anemia in younger patients with newly diagnosed acute myeloid leukemia. Studying samples of tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to Fanconi anemia in patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify children with newly diagnosed acute myeloid leukemia (AML) treated on COG-2961 and COG-AAML03P1 who are at high risk of having de novo Fanconi anemia.

II. Procure diagnostic samples from the COG AML Biology Repository and identify Fanconi anemia patients using western blot techniques.

OUTLINE:

Previously collected cryopreserved cells are analyzed via western blot to identify patients with Fanconi anemia.

ELIGIBILITY:
Inclusion Criteria:

* Treated on COG-2961 or COG-AAML03P1
* At high risk of having Fanconi anemia, defined as meeting one the following groups of clinical criteria:

  * Group 1: Prolonged neutropenia after induction, severe regimen-related toxicity (mucositis, veno-occlusive disease, end-organ damage)
  * Group 2: Early non-relapse death (induction, consolidation)
  * Group 3: Small-for-weight, secondary malignancies

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients treated on trials COG-2961 or COG-AAML03P1. Also patients at high risk of having Fanconi anemia meeting other criteria.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Identification of children at high risk of having Fanconi anemia | Up to 5 months
Identification of Fanconi anemia patients | Up to 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Monica Thakar, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States